CLINICAL TRIAL: NCT05060588
Title: The Effect of Sacubitril/Valsartan Versus Valsartan on the Short-term Prognosis of Hypertensive Patients With Acute Myocardial Infarction
Brief Title: Sacubitril/Valsartan Versus Valsartan for Hypertensive Patients With Acute Myocardial Infarction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qingdao Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Sacu-HPT
Record Dates: First submitted 2021-09-13; First posted 2021-09-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Myocardial Infarction; Hypertension
Keywords: Sacubitril/Valsartan; Valsartan; Myocardial Infarction; Hypertension
MeSH Terms: conditions — Myocardial Infarction; Hypertension | interventions — sacubitril; Valsartan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sacubitril/Valsartan (Experimental): Sacubitril/Valsartan 24/26 mg once every 12 hours for 6 months
  Interventions: Drug: Sacubitril/Valsartan 49/51mg/Tab
- Valsartan (Active Comparator): 1 tablet of Valsartan every 24 hours for 6 months
  Interventions: Drug: Valsartan 80mg/Tab

INTERVENTIONS:
Drug: Sacubitril/Valsartan 49/51mg/Tab — patients who meet the inclusion criteria are randomized to receive Sacubitril/Valsartan 24/26 mg once every 12 hours for 6 months
  Other Names: Sacubitril/Valsartan Group
  Arms: Sacubitril/Valsartan
Drug: Valsartan 80mg/Tab — Patients who meet the inclusion criteria are randomized to receive valsartan one tablet every 24 hours for 6 months.
  Other Names: Valsartan Group
  Arms: Valsartan

SUMMARY:
Studies have demonstrated that the early initiation of ACEI/ARB to patients with acute myocardial infarction is beneficial, especially in patients combined with reduced LVEF or mild-moderate heart failure. Therefore, ACEI/ARB is a traditional treatment for patients post-infarction. Recent clinical trials have demonstrated that Sacubitril/Valsartan is more beneficial than Ramipril to patients post-PCI.Besides, Sacubitril/Valsartan is also effective for essential hypertension.This study aims to assess the effect of Sacubitril/Valsartan on short-term prognosis in hypertensive patients with acute myocardial infarction compared against Valsartan.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with new-onset MI, either STEMI or NSTEMI, according to the fourth universal definition of MI (Thygesen et al. 2019), disease onset within 7 days.
2. Patients are previously diagnosed with essential hypertension or newly diagnosed with essential hypertension.
3. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and the protocol.

Exclusion Criteria:

1. Patients with severe renal dysfunction. (GFR<60mmol/L).
2. Patients who have recently undergone immunosuppressive therapy.
3. Patients who are known to be allergic to Sacubitril/Valsartan and Valsartan.
4. Patients who are hemodynamically unstable.
5. Chronic symptomatic heart failure within the last year and known reduced ejection fraction (LVEF≤40 %).
6. Severe hepatic impairment (Child-Pugh class C) at the time of inclusion into the trial.
7. Any non-CV condition, such as active malignancy requiring treatment at the time of screening, or severe diseases with a life expectancy of fewer than two years based on the investigator´s clinical judgment.
8. Currently on treatment with Sacubitril/Valsartan or an ACEI/ARB.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Rate of MACE events no.1 by phone calls and questionnaires | 6 months
  To assess the rate of myocardial infarction in post-infarction patients during the study follow-up.
Rate of MACE events No.2 by phone calls and questionnaires | 6 months
  To assess the rate of stroke in patients post-MI during the follow up period
Rate of MACE events No.3 phone calls and questionnaires | 6 months
  To assess the rate of death from cardiovascular causes during the follow up time

SECONDARY OUTCOMES:
Left ventricular ejection fraction(LVEF) by echocardiography | 6 months
  Evaluate baseline left ventricular ejection fraction (LVEF)in post-infarct patients and 6 months of treatment.
Rate of post infarction angina by following up in the clinic | 6 months
  Evaluate the Effect of Sacubitril/Valsartan versus Valsartan on the development of post-infarction angina.
The rate of heart failure occurrence by following up in the clinic | 6 months
  Assess the occurence of heart failure during the study follow-up.
Left ventricular end-diastolic volume(LVEDV) by echocardiography | 6 months
  Evaluate the baseline LVEDV in post-infarct patients and 6 months of treatment using echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Jun Teng, MD, Study Director — Qingdao Central Hospital
Locations (1):
- Mengmei Li, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No